CLINICAL TRIAL: NCT05770726
Title: The Comparison of the Adjuvant Effect of Probiotics Between Delivery Via Colonoscopic Spray and Oral Administration in Patients With Clostridioides Difficile Colitis Receiving Vancomycin Treatment
Brief Title: Probiotics Administration Via Colonoscopic Spray and Oral Administration in CDAD Patients
Acronym: CDAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-111-052
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-01

CONDITIONS: Diarrhea Infectious
Keywords: Clostridioides difficile colitis
MeSH Terms: conditions — Dysentery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotics-spray (PS) group (Active Comparator): In the PS group, the colonoscopic prescription of 10 grams of probiotics powder is performed once on one of the first three days (D0-D3).
  Interventions: Dietary Supplement: Probiotics administration
- probiotics-oral (PO) group (Active Comparator): In the PO group, we will prescribe oral probiotics 2 capsules once per day for 5 days (a total of 10 grams) as adjunctive treatment during the first five days (D0-D4).
  Interventions: Dietary Supplement: Probiotics administration

INTERVENTIONS:
Dietary Supplement: Probiotics administration — A total of 10 grams of probiotics was administered in both group, but the routes were different. One group were per colonoscopic spray, and the other was per oral.

SUMMARY:
Clostridioides difficile (C. difficile) colitis is a common hospital-acquired disease, which increases hospitalization length and the mortality rate. Moreover, refractory or recurrent C. difficile colitis is an emerging disease. The tapering course of oral vancomycin or oral fidaxomicin is current standard treatment for refractory or recurrent C. difficile colitis. Fecal microbiota transplantation (FMT) is an alternative one. However, the tapering course of oral vancomycin needs a 6- to 12-week duration, fidaxomicin is expensive, and FMT is not available in every hospital; therefore, it is needed to develop a new treatment. Evidence has shown that the disturbance with reduced diversity of intestinal microbiota may lead to refractory C. difficile colitis. Besides fecal microbiota transplantation, probiotics administration can also correct the disturbed intestinal microbiota. However, inconsistent efficacy of probiotic administration was reported, which may be attributed to the interference by the gastric acid. Precise delivery of probiotics into the colon by colonoscopy can avoid the destruction by gastric acid, with which a better treatment efficacy is expected. The best regimen for C. difficile colitis should be the one which succeeds on the first attempt. Therefore, this study is aimed toward validating the efficacy and safety of the colonoscopic probiotics-spray.

Patients diagnosed with C. colitis will be enrolled. All patients will accept the standard treatment of oral vancomycin for 14 days. As an adjuvant probiotic administration at the same time, enrolled patients will be randomly assigned to the probiotics-spray (PS) group and the probiotics-oral (PO) group, respectively. The patients in the PS group will receive colonoscopic spray of probiotics once, while the patients in the PO group will receive the same dosage of oral probiotics divided into 5 days. This study will compare the difference in fecal microbiota changes between the colonoscopic probiotics-spray group and the probiotics-oral group. Moreover, this study will evaluate the efficacy and safety between the colonoscopic probiotics-spray and probiotics-oral in patients with C. difficile colitis.

DETAILED DESCRIPTION:
Refractory or recurrent C. difficile colitis is an emerging disease. The tapering course of oral vancomycin or oral fidaxomicin is current standard treatment for refractory or recurrent C. difficile colitis.FMT is an alternative treatment. Nevertheless, the tapering course of oral vancomycin needs a 6- to 12-week duration, fidaxomicin is expensive, and FMT is not available in many hospitals. Therefore, we need a method which is effective for patients and available for clinicians.

The disturbance with reduced diversity of intestinal microbiota may lead to refractory or recurrent C. difficile colitis. Moreover, the probiotics administration can correct the disturbed intestinal microbiota. However, inconsistent efficacy of probiotic administration was reported, which may be attributed to the interference by the gastric acid. There is no exact estimation for the amounts of probiotics in the colon after oral administration. Moreover, there is no study which is conducted to compare the efficiency of probiotics between direct spray via colonoscopy and oral administration. It will be novel to study such issue. If the amounts of probiotics which is delivered directly via colonoscopy and the clinical efficacy are similar to those by FMT, colonoscopic probiotics-spray will replace FMT in clinical practice.

FMT can correct the disturbed intestinal microbiota. The estimated bacteria of human wet stool are 1011 per gram. The amount of stool for FMT is ~30 to 100 grams; thus, ~1012 to 1013 bacteria will be transplanted in an FMT procedure. In this project, we will transplant ~2x1011 probiotics into the colon by the colonoscopic spray. Therefore, we believe that colonoscopic spray of probiotics will have similar amounts of bacteria transplanted with FMT but be more efficient than oral probiotics administration.

Probiotics use may have adverse events. There are few studies and case reports which recorded that the administered probiotic was isolated from sterile sites, such as bacteremia. Thus, the safety issue of this study will focus on the adverse events, bacteremia and sepsis.

It will be novel to conduct the study to compare the efficacy and safety of probiotics which are delivered directly via colonoscopy and oral administration. If it works, colonoscopic probiotics spray will replace FMT in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 20 years who are diagnosed with C. difficile colitis

Exclusion Criteria:

* patients are diagnosed with colitis because of other etiologies, such as intestinal Behçet's disease, amoeba or parasitic colitis, Salmonella colitis, lymphoma, E. coli colitis, cytomegalovirus colitis, ischemic colitis, sigmoid-colon cancer, inflammatory bowel diseases (ulcerative colitis or Crohn's disease), solitary rectal ulcer syndrome, radiation colitis
* patients who have contraindications for colonoscopy, including declining or refusal to cooperate
* unstable vital signs
* a diagnosis or highly suspicion of colon rupture
* a high-risk situation for colon perforation such as acute diverticulitis
* toxic megacolon, etc.
* acute myocardial infarct

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of difference in fecal microbiota change, including probiotics, between the colonoscopic probiotics-spray and probiotics-oral and before and after probiotics use either by colonoscopic probiotics-spray or probiotics-oral | 5 days
  All patients will be monitored for 30 days after diagnosis of C. difficile colitis. The primary endpoint is the comparison of the perseverance of fecal microbiota and metabolites. We will compare the microbiota by sequencing 16S rRNA, measured as percentage abundance per microbial species and differences in percentage abundance between the PS group and PO group in Day 0 and Day 5. We will also compare the relative abundance of C. difficile and target probiotics between the two study groups, such as Lactobacillus acidophilus, Bifidobacterium bifidum, Streptococcus thermophilus, or others.

SECONDARY OUTCOMES:
The rate of resolution of C. difficile colitis | 30 days
  the resolution time of diarrhea and bloody stool
Hospitalization length | 30 days
  the total hospitalization length
The rate of recurrence of C. difficile colitis | 30 days
  the recurrence of C. difficile colitis
The rate of mortality events | 30 days
  all-cause mortality
The rate of adverse events | 30 days
  adverse events from probiotics, including probiotics bacteremia and sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh-Chien Chiang, M.D., Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Other (Non U.s.), Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing after the study completed and the paper published

REFERENCES:
- [Result] McDonald LC, Gerding DN, Johnson S, Bakken JS, Carroll KC, Coffin SE, Dubberke ER, Garey KW, Gould CV, Kelly C, Loo V, Shaklee Sammons J, Sandora TJ, Wilcox MH. Clinical Practice Guidelines for Clostridium difficile Infection in Adults and Children: 2017 Update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA). Clin Infect Dis. 2018 Mar 19;66(7):e1-e48. doi: 10.1093/cid/cix1085. PMID 29462280
- [Result] Bagdasarian N, Rao K, Malani PN. Diagnosis and treatment of Clostridium difficile in adults: a systematic review. JAMA. 2015 Jan 27;313(4):398-408. doi: 10.1001/jama.2014.17103. PMID 25626036
- [Result] Kelly CP, LaMont JT. Clostridium difficile--more difficult than ever. N Engl J Med. 2008 Oct 30;359(18):1932-40. doi: 10.1056/NEJMra0707500. No abstract available. PMID 18971494
- [Result] Kelly CR, Fischer M, Allegretti JR, LaPlante K, Stewart DB, Limketkai BN, Stollman NH. ACG Clinical Guidelines: Prevention, Diagnosis, and Treatment of Clostridioides difficile Infections. Am J Gastroenterol. 2021 Jun 1;116(6):1124-1147. doi: 10.14309/ajg.0000000000001278. PMID 34003176
- [Result] Goodhand JR, Alazawi W, Rampton DS. Systematic review: Clostridium difficile and inflammatory bowel disease. Aliment Pharmacol Ther. 2011 Feb;33(4):428-41. doi: 10.1111/j.1365-2036.2010.04548.x. Epub 2010 Dec 30. PMID 21198703
- [Result] Chang JY, Antonopoulos DA, Kalra A, Tonelli A, Khalife WT, Schmidt TM, Young VB. Decreased diversity of the fecal Microbiome in recurrent Clostridium difficile-associated diarrhea. J Infect Dis. 2008 Feb 1;197(3):435-8. doi: 10.1086/525047. PMID 18199029
- [Result] Mullish BH, Quraishi MN, Segal JP, McCune VL, Baxter M, Marsden GL, Moore DJ, Colville A, Bhala N, Iqbal TH, Settle C, Kontkowski G, Hart AL, Hawkey PM, Goldenberg SD, Williams HRT. The use of faecal microbiota transplant as treatment for recurrent or refractory Clostridium difficile infection and other potential indications: joint British Society of Gastroenterology (BSG) and Healthcare Infection Society (HIS) guidelines. Gut. 2018 Nov;67(11):1920-1941. doi: 10.1136/gutjnl-2018-316818. Epub 2018 Aug 28. PMID 30154172
- [Result] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Result] Hemarajata P, Versalovic J. Effects of probiotics on gut microbiota: mechanisms of intestinal immunomodulation and neuromodulation. Therap Adv Gastroenterol. 2013 Jan;6(1):39-51. doi: 10.1177/1756283X12459294. PMID 23320049
- [Result] Hempel S, Newberry SJ, Maher AR, Wang Z, Miles JN, Shanman R, Johnsen B, Shekelle PG. Probiotics for the prevention and treatment of antibiotic-associated diarrhea: a systematic review and meta-analysis. JAMA. 2012 May 9;307(18):1959-69. doi: 10.1001/jama.2012.3507. PMID 22570464
- [Result] Phanchana M, Harnvoravongchai P, Wongkuna S, Phetruen T, Phothichaisri W, Panturat S, Pipatthana M, Charoensutthivarakul S, Chankhamhaengdecha S, Janvilisri T. Frontiers in antibiotic alternatives for Clostridioides difficile infection. World J Gastroenterol. 2021 Nov 14;27(42):7210-7232. doi: 10.3748/wjg.v27.i42.7210. PMID 34876784
- [Result] Pillai A, Nelson R. Probiotics for treatment of Clostridium difficile-associated colitis in adults. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD004611. doi: 10.1002/14651858.CD004611.pub2. PMID 18254055
- [Result] Corcoran BM, Stanton C, Fitzgerald GF, Ross RP. Survival of probiotic lactobacilli in acidic environments is enhanced in the presence of metabolizable sugars. Appl Environ Microbiol. 2005 Jun;71(6):3060-7. doi: 10.1128/AEM.71.6.3060-3067.2005. PMID 15933002
- [Result] Han S, Lu Y, Xie J, Fei Y, Zheng G, Wang Z, Liu J, Lv L, Ling Z, Berglund B, Yao M, Li L. Probiotic Gastrointestinal Transit and Colonization After Oral Administration: A Long Journey. Front Cell Infect Microbiol. 2021 Mar 10;11:609722. doi: 10.3389/fcimb.2021.609722. eCollection 2021. PMID 33791234
- [Result] Staley C, Halaweish H, Graiziger C, Hamilton MJ, Kabage AJ, Galdys AL, Vaughn BP, Vantanasiri K, Suryanarayanan R, Sadowsky MJ, Khoruts A. Lower endoscopic delivery of freeze-dried intestinal microbiota results in more rapid and efficient engraftment than oral administration. Sci Rep. 2021 Feb 25;11(1):4519. doi: 10.1038/s41598-021-84152-6. PMID 33633264
- [Result] Honda H, Dubberke ER. Clostridium difficile infection: a re-emerging threat. Mo Med. 2009 Jul-Aug;106(4):287-91. PMID 19753922
- [Result] Wu KS, Syue LS, Cheng A, Yen TY, Chen HM, Chiu YH, Hsu YL, Chiu CH, Su TY, Tsai WL, Chen WY, Huang CH, Hung HM, Huang LJ, Kuo HJ, Lin PC, Yang CH, Hong PL, Lee SS, Chen YS, Liu YC, Huang LM; Infectious Diseases Society of Taiwan; Medical Foundation in Memory of Dr. Deh-Lin Cheng; Foundation of Professor Wei-Chuan Hsieh for Infectious Diseases Research and Education; CY Lee's Research Foundation for Pediatric Infectious Diseases and Vaccines; 5th Guidelines Recommendations for Evidence-based Antimicrobial agents use in Taiwan (GREAT) working group. Recommendations and guidelines for the treatment of Clostridioides difficile infection in Taiwan. J Microbiol Immunol Infect. 2020 Apr;53(2):191-208. doi: 10.1016/j.jmii.2020.02.002. Epub 2020 Feb 14. PMID 32169531
- [Result] Surawicz CM, Alexander J. Treatment of refractory and recurrent Clostridium difficile infection. Nat Rev Gastroenterol Hepatol. 2011 Jun;8(6):330-9. doi: 10.1038/nrgastro.2011.59. Epub 2011 Apr 19. PMID 21502971
- [Result] Chilton CH, Pickering DS, Freeman J. Microbiologic factors affecting Clostridium difficile recurrence. Clin Microbiol Infect. 2018 May;24(5):476-482. doi: 10.1016/j.cmi.2017.11.017. Epub 2017 Dec 5. PMID 29208562
- [Result] Ma C, Wasti S, Huang S, Zhang Z, Mishra R, Jiang S, You Z, Wu Y, Chang H, Wang Y, Huo D, Li C, Sun Z, Sun Z, Zhang J. The gut microbiome stability is altered by probiotic ingestion and improved by the continuous supplementation of galactooligosaccharide. Gut Microbes. 2020 Nov 9;12(1):1785252. doi: 10.1080/19490976.2020.1785252. Epub 2020 Jul 14. PMID 32663059
- [Result] Dodoo CC, Wang J, Basit AW, Stapleton P, Gaisford S. Targeted delivery of probiotics to enhance gastrointestinal stability and intestinal colonisation. Int J Pharm. 2017 Sep 15;530(1-2):224-229. doi: 10.1016/j.ijpharm.2017.07.068. Epub 2017 Jul 29. PMID 28764983
- [Result] Bojanova DP, Bordenstein SR. Fecal Transplants: What Is Being Transferred? PLoS Biol. 2016 Jul 12;14(7):e1002503. doi: 10.1371/journal.pbio.1002503. eCollection 2016 Jul. PMID 27404502
- [Result] Ledoux D, Labombardi VJ, Karter D. Lactobacillus acidophilus bacteraemia after use of a probiotic in a patient with AIDS and Hodgkin's disease. Int J STD AIDS. 2006 Apr;17(4):280-2. doi: 10.1258/095646206776253507. PMID 16595054
- [Result] Johnstone J, Meade M, Lauzier F, Marshall J, Duan E, Dionne J, Arabi YM, Heels-Ansdell D, Thabane L, Lamarche D, Surette M, Zytaruk N, Mehta S, Dodek P, McIntyre L, English S, Rochwerg B, Karachi T, Henderson W, Wood G, Ovakim D, Herridge M, Granton J, Wilcox ME, Goffi A, Stelfox HT, Niven D, Muscedere J, Lamontagne F, D'Aragon F, St-Arnaud C, Ball I, Nagpal D, Girard M, Aslanian P, Charbonney E, Williamson D, Sligl W, Friedrich J, Adhikari NK, Marquis F, Archambault P, Khwaja K, Kristof A, Kutsogiannis J, Zarychanski R, Paunovic B, Reeve B, Lellouche F, Hosek P, Tsang J, Binnie A, Trop S, Loubani O, Hall R, Cirone R, Reynolds S, Lysecki P, Golan E, Cartin-Ceba R, Taylor R, Cook D; Prevention of Severe Pneumonia and Endotracheal Colonization Trial (PROSPECT) Investigators and the Canadian Critical Care Trials Group. Effect of Probiotics on Incident Ventilator-Associated Pneumonia in Critically Ill Patients: A Randomized Clinical Trial. JAMA. 2021 Sep 21;326(11):1024-1033. doi: 10.1001/jama.2021.13355. PMID 34546300
- [Result] Georgieva R, Yocheva L, Tserovska L, Zhelezova G, Stefanova N, Atanasova A, Danguleva A, Ivanova G, Karapetkov N, Rumyan N, Karaivanova E. Antimicrobial activity and antibiotic susceptibility of Lactobacillus and Bifidobacterium spp. intended for use as starter and probiotic cultures. Biotechnol Biotechnol Equip. 2015 Jan 2;29(1):84-91. doi: 10.1080/13102818.2014.987450. Epub 2014 Dec 11. PMID 26019620